CLINICAL TRIAL: NCT00588068
Title: Molecular Characterization of Neuroblastic Tumor: Correlation With Clinical Outcome
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Southern Illinois University (Other); Spanish National Cancer Center (Unknown); St. Jude Children's Research Hospital (Other); Washington University School of Medicine (Other); University of Texas (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 00-109
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Neuroblastoma
Keywords: Adrenal Gland; No stage requirement
MeSH Terms: conditions — Neuroblastoma | interventions — Tumor Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor, marrow and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Tumor and Marrow Markers
  Interventions: Other: Tumor and Marrow Markers

INTERVENTIONS:
Other: Tumor and Marrow Markers — Tumor and Marrow Markers

SUMMARY:
The purpose of this study is to find out the genetic and biochemical makeup of your neuroblastic tumor, which influences its aggressiveness and the suitable therapy. These research studies include surface marker analysis, cytogenetics, cancer genes,genome sequencing, tumor growth-related genes and tumor growth in test tubes. Your blood, marrow, and hematopoietic stem cell samples will also be tested for tumors or leukemia cells, and your serum tested for anti-tumor antibodies.

DETAILED DESCRIPTION:
To collect tumor, marrow specimens prospectively to study the molecular-genetic makeup of individual neuroblastic tumor and its metastasis by blood and marrow, and to correlate these findings with clinical outcome, and to relate the signaling circuitry of neuroblastic tumors to that of embryonic neuroectodermal cells. .

ELIGIBILITY:
Inclusion Criteria:

* Neuroblastic tumors diagnosed in accordance with the International Neuroblastoma Staging System

OR

* Clinically suspected neuroblastic tumors.

PK DRAW INCLUSION CRITERIA (FOR PK DRAWS ONLY):

PK Draw Inclusion Criteria

* Patients who receive naxitamab as part of their standard of care

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be offered participation in this study by their attending oncologist in the Department of Pediatrics at Memorial Sloan Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 2070 (Estimated)
Dates: Start 2000-09-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To study the molecular-genetic makeup and metastasis of neuroblastic tumors. | 2 years
  Before surgery a maximum of 5 blood drawings (20-30 ml) will be performed per year (at least one month apart) per patient

SECONDARY OUTCOMES:
To study the correlation of these biologic markers with clinical outcome. | 2 years
  Before surgery and a maximum of 5 blood drawings (20-30 ml) will be performed per year (at least one month apart) per patient
To relate neuroblastic tumor and embryonic neuroectodermal cell circuitry. | 2 years
  Up to six fetal adrenal samples will be obtained (without patient identifiers) from gestational week 20, when neuroblasts are present and thought to be differentiating within the fetal adrenal gland.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong Cheung, M.D., Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Felix CA, Slater DJ, Davenport JW, Yu X, Gregory BD, Li MM, Rappaport EF, Cheung NV. KMT2A-MAML2 rearrangement emerged and regressed during neuroblastoma therapy without leukemia after 12.8-year follow-up. Pediatr Blood Cancer. 2022 Jan;69(1):e29344. doi: 10.1002/pbc.29344. Epub 2021 Sep 22. PMID 34550633
- [Derived] Cheung NK, Zhang J, Lu C, Parker M, Bahrami A, Tickoo SK, Heguy A, Pappo AS, Federico S, Dalton J, Cheung IY, Ding L, Fulton R, Wang J, Chen X, Becksfort J, Wu J, Billups CA, Ellison D, Mardis ER, Wilson RK, Downing JR, Dyer MA; St Jude Children's Research Hospital-Washington University Pediatric Cancer Genome Project. Association of age at diagnosis and genetic mutations in patients with neuroblastoma. JAMA. 2012 Mar 14;307(10):1062-71. doi: 10.1001/jama.2012.228. PMID 22416102
- See also: Memorial Sloan Kettering Cancer Center website — http://www.mskcc.org